CLINICAL TRIAL: NCT05363644
Title: Treatment Protocol With BioDFence® G3 For Full Nerve-Sparing Robotic-Assisted Radical Prostatectomy: A Prospective Open Label Single-Center Study
Brief Title: BioDFence® G3 For Full Nerve-Sparing Robotic-Assisted Radical Prostatectomy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was withdrawn due to lack of funding
Sponsor: AdventHealth (Other)
Collaborators: Integra LifeSciences Corporation (Industry)
Responsible Party: Principal Investigator, Vipul Patel, MD, Dr. Vipul R. Patel, AdventHealth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1803935
Record Dates: First submitted 2022-04-25; First posted 2022-05-06 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Prostate Cancer; Prostatectomy; Erectile Dysfunction Following Radical Prostatectomy; Incontinence, Urinary
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: All of the patients will be recruited from patients seen in the principal investigator's (PI's) hospital and practice. The offer to participate will be extended to all eligible subjects for the importance of a representative sample.
  No women, children or prisoners will be enrolled in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single Arm Study Group (Experimental): Placement of a sheet of BioDFence G3 to the neurovascular bundle.
  Interventions: Biological: BioDFence G3

INTERVENTIONS:
Biological: BioDFence G3 — Placement of a sheet of BioDFence® G3 will be applied to the neurovascular bundle on participants undergoing an elective Full Nerve Sparing Radical Prostatectomy for primary treatment of prostate cancer.

SUMMARY:
The purpose of this study is to assess functional outcomes post operatively after the use of BioDFence® G3 during robotic radical prostatectomy.

DETAILED DESCRIPTION:
The purpose of this study is to build on our experience of amniotic membrane use in Robotic Assisted Radical Prostatectomy for prostate cancer, we aim to evaluate clinical outcomes related to the use of BioDFence® G3; a tri-layered amniotic membrane. BioDFence® G3 is regulated by the FDA as a 361 HCT/P for use from head to toe as a tissue barrier for soft tissue repair and as a wound covering.

For the purpose of this study BioDFence® G3 will be placed on the neurovascular bundles by the surgeon during the robotic assisted radical prostatectomy procedure that the participant has elected as their primary treatment for prostate cancer. The potential benefits that will be assessed are an earlier return of potency after surgery as evidenced by The Sexual Health Inventory for Men (SHIM) questionnaire score and self-reported sexual function and secondarily looking at continence outcomes measured by The American Urological Association (AUA) questionnaire form and self-reported urinary function.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects between the ages 40-70.
2. Primary diagnosis of prostate cancer requiring surgical intervention
3. Have a willingness to comply with follow-up requirements.
4. Have ability to provide full written consent.
5. Primary diagnosis of untreated with clinically localized prostate cancer with Gleason score of 6, or 7.
6. Planned elective radical prostatectomy with bilateral full nerve sparing technique.
7. Patients who currently have a pre-operative SHIM > 19

Exclusion Criteria:

1. Has signs or symptoms of any other disease which could result in allograft failure or has experienced graft failure in the past.
2. Has any condition(s), which seriously compromises the subject's ability to participate in this study or has a known history of poor adherence with medical treatment.
3. Has comorbid conditions that can be confused with or can exacerbate the condition of erectile dysfunction, including:

   1. Diabetes Type I or Type II
   2. Advanced atherosclerotic vascular disease
4. Is unable to sign or understand informed consent.
5. Is unable to comply with penile rehabilitation, including oral 5-phosphodiesterase inhibitor.
6. Has a documented medical history of drug or alcohol abuse within last 12 months.
7. Has autoimmune disease or a known history of having Acquired Immunodeficiency Syndrome (AIDS) or HIV.
8. Known sensitivity to glutaraldehyde or ethanol.
9. Patients with a history of more than two weeks treatment with immuno-suppressants (including systemic corticosteroids), cytotoxic chemotherapy within one month prior to initial screening, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study.
10. Has had prior hormonal therapy such as Lupron or oral anti-androgens.
11. Living outside of United States
12. Partial nerve sparing technique used during Radical Prostatectomy

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to potency | 14 days to 12 months post prostatectomy
  Outcome measured by the Sexual Health Inventory for Men (SHIM) score and patient reported potency erectile function score.

SECONDARY OUTCOMES:
Time to continence | 14 days to 12 months post prostatectomy
  Outcome measured by the American Urological Association (AUA ) score and patient reported number of urinary sanitation pads used daily.

CONTACTS AND LOCATIONS:
Overall Officials: Vipul R Patel, MD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth, Celebration, Florida, United States

IPD SHARING:
Plan to Share IPD: No
De-identified information may be utilized in teachings and/or publication as it related to this research.

REFERENCES:
- [Background] Shrader-Bogen CL, Kjellberg JL, McPherson CP, Murray CL. Quality of life and treatment outcomes: prostate carcinoma patients' perspectives after prostatectomy or radiation therapy. Cancer. 1997 May 15;79(10):1977-86. doi: 10.1002/(sici)1097-0142(19970515)79:103.0.co;2-r. PMID 9149026
- [Background] Walsh PC. Patient-reported urinary continence and sexual function after anatomic radical prostatectomy. J Urol. 2000 Jul;164(1):242. No abstract available. PMID 10896513
- [Background] Catalona WJ, Carvalhal GF, Mager DE, Smith DS. Potency, continence and complication rates in 1,870 consecutive radical retropubic prostatectomies. J Urol. 1999 Aug;162(2):433-8. PMID 10411052
- [Background] Rabbani F, Stapleton AM, Kattan MW, Wheeler TM, Scardino PT. Factors predicting recovery of erections after radical prostatectomy. J Urol. 2000 Dec;164(6):1929-34. PMID 11061884
- [Background] Stanford JL, Feng Z, Hamilton AS, Gilliland FD, Stephenson RA, Eley JW, Albertsen PC, Harlan LC, Potosky AL. Urinary and sexual function after radical prostatectomy for clinically localized prostate cancer: the Prostate Cancer Outcomes Study. JAMA. 2000 Jan 19;283(3):354-60. doi: 10.1001/jama.283.3.354. PMID 10647798
- [Background] Patel VR, Samavedi S, Bates AS, Kumar A, Coelho R, Rocco B, Palmer K. Dehydrated Human Amnion/Chorion Membrane Allograft Nerve Wrap Around the Prostatic Neurovascular Bundle Accelerates Early Return to Continence and Potency Following Robot-assisted Radical Prostatectomy: Propensity Score-matched Analysis. Eur Urol. 2015 Jun;67(6):977-980. doi: 10.1016/j.eururo.2015.01.012. Epub 2015 Jan 19. PMID 25613153
- [Background] Magatti M, De Munari S, Vertua E, Parolini O. Amniotic membrane-derived cells inhibit proliferation of cancer cell lines by inducing cell cycle arrest. J Cell Mol Med. 2012 Sep;16(9):2208-18. doi: 10.1111/j.1582-4934.2012.01531.x. PMID 22260183
- [Background] Wang TM. [Evaluation of the use of human amnion as a biological dressing]. Zhonghua Zheng Xing Shao Shang Wai Ke Za Zhi. 1986 Dec;2(4):282-3. No abstract available. Chinese. PMID 3151296
- [Background] DANFORTH D, HULL RW. The microscopic anatomy of the fetal membranes with particular reference to the detailed structure of the amnion. Am J Obstet Gynecol. 1958 Mar;75(3):536-47; discussion 548-50. doi: 10.1016/0002-9378(58)90610-0. No abstract available. PMID 13508744
- [Background] Walsh PC. Nerve grafts are rarely necessary and are unlikely to improve sexual function in men undergoing anatomic radical prostatectomy. Urology. 2001 Jun;57(6):1020-4. doi: 10.1016/s0090-4295(01)00987-6. No abstract available. PMID 11377297
- [Background] Menon M, Kaul S, Bhandari A, Shrivastava A, Tewari A, Hemal A. Potency following robotic radical prostatectomy: a questionnaire based analysis of outcomes after conventional nerve sparing and prostatic fascia sparing techniques. J Urol. 2005 Dec;174(6):2291-6, discussion 2296. doi: 10.1097/01.ju.0000181825.54480.eb. PMID 16280816